CLINICAL TRIAL: NCT06228755
Title: Scaling-Up Integrative Pain Management in Federally-Qualified Health Centers
Brief Title: MAGIC Study: More Access to Group Integrative Care
Acronym: MAGIC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-2481; 5K01AT011578-02 (NIH)
Record Dates: First submitted 2024-01-16; First posted 2024-01-29 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training, Coaching, and Orientation (Experimental): Clinic personnel will receive training for delivering integrative medicine group visits (IMGV) and ongoing coaching in delivering IMGV for patients with chronic pain. Clinic patients will participate in orientation and the 9-week IMGV.
  Interventions: Behavioral: Integrative Medicine Group Visit; Other: Implementation Strategies

INTERVENTIONS:
Behavioral: Integrative Medicine Group Visit — Integrative Medicine Group Visit (IMGV) is a 9-week group visit series co-facilitated by a billing primary care provider and a trained co-facilitator (such as a behavioral health provider, mindfulness instructor, or yoga teacher). The IMGV will be delivered virtually over a secure telehealth platform for 2 hours weekly. The IMGV curriculum focuses on principles of mindfulness-based stress reduction, and includes patient education on pain, insomnia, nutrition, yoga, depression, self-massage, and self-acupressure.
  Other Names: IMGV
Other: Implementation Strategies — Package includes:
  * Patient strategies will include an orientation session to introduce patients to the IMGV model.
  * Provider strategies include training in delivery of IMGV with continuing education credits. Training may be delivered on-line or in-person. Ongoing coaching in the first year of IMGV implementation will also be offered to providers leading IMGV, to increase self-efficacy to deliver the curriculum, and enhance fidelity.
  Other Names: Implementation Strategies Package

SUMMARY:
Chronic pain impacts about 20% of US Adults. Though non-pharmacologic, integrative pain management therapies are now considered first-line treatment by clinical guidelines, these therapies are still rarely covered by health insurance and therefore inaccessible to lower-income individuals. The Integrative Medical Group Visit (IMGV) program was developed to offer low-income, diverse patients with chronic pain an introduction to integrative pain management approaches, through a model that is covered by health insurance under existing billing codes. An initial pragmatic randomized control trial found that IMGV led to significant improvement in mental health related quality of life and lower use of high-cost care. However, there has been little research investigating the implementation of IMGV, and none in Federally-Qualified Health Centers (FQHCs), where the program was initially designed to be implemented. In this study, the investigators test strategies to implement IMGV in FQHCs, including training and coaching clinic staff, and measure the effectiveness of the IMGV on health outcomes for patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Staff and clinicians at each clinic who are involved in implementation of the IMGV.
* Only patients who have enrolled in the Integrative medical group visit (IMGV) programs for patients with chronic pain at their Federally Qualified Health Center will be eligible for enrollment in the study. Physicians at each clinical site will determine enrollment criteria for their IMGV program specific to their clinical site--patients who are enrolled in the program will then be invited to participate in the research study.

Exclusion Criteria:

* All staff, clinicians, and patients who are not involved in the IMGV at the specific clinical sites are excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Reach: Total Patients Reached | through study completion, a total of up to 3 years
  Number of patients who enroll in IMGV at each clinical site.
Reach: Race of Patients Reached | through study completion, a total of up to 3 years
  Race of patients who enroll in IMGV at each clinical site.
Reach: Ethnicity of Patients Reached | through study completion, a total of up to 3 years
  Ethnicity of patients who enroll in IMGV at each clinical site.
Reach: Gender of Patients Reached | through study completion, a total of up to 3 years
  Gender of patients who enroll in IMGV at each clinical site.
Reach: Age of Patients Reached | through study completion, a total of up to 3 years
  Age of patients who enroll in IMGV at each clinical site.
Adoption | through study completion, a total of up to 3 years
  Number of clinic staff willing to form an implementation team to participate in delivering and implementing the IMGV at each clinical site.
Acceptability: Patients | within 1 month of final IMGV session participation, approximately 10 weeks
  Number of patients who perceive the IMGV to be acceptable based on qualitative data analysis.
Acceptability: Clinic Personnel | within 1 month of final IMGV session participation, approximately 10 weeks
  Number of clinic personnel who perceive the implementation of IMGV to be acceptable based on qualitative data analysis.
Cost: Patient Perspective | within 1 month of final IMGV session participation, approximately 10 weeks
  Total cost of participation in the IMGV from the perspective of patients (ie total cost of time, accessing technology, childcare, out-of-pocket costs).
Cost: Clinic Perspective | within 1 month of final IMGV session participation, approximately 10 weeks
  Total cost of implementation in the IMGV from the perspective of the clinic (ie total cost of staff time to implement the program, material costs).
Fidelity | Through completion of IMGV delivery, a total of up to two years
  Score on the Integrative Medical Group Visit (IMGV) Fidelity rating scale, measuring the extent to which core functions of the IMGV were delivered as intended by the clinic personnel. The scale includes 5 questions using a 0-3 point scale. Questions measure the constructs: fostering a safe and positive environment, fostering social support through the group, providing evidence-based medical advice, fostering collaboration, and providing access to integrative therapy experiential practice. Total range is from 0-15 with 0 representing the lowest and 15 representing the highest possible fidelity.
Maintenance: 6 months | Six months after the first IMGV session at clinic
  Number of IMGV sessions held at the clinic at 6 months since the first IMGV session at that clinic.
Maintenance: 12 months | Twelve months after the first IMGV session at clinic
  Number of IMGV sessions held at the clinic at 12 months since the first IMGV session at that clinic.

SECONDARY OUTCOMES:
Change in Physical Function | Pre-assessments will be conducted within 4 weeks of the first IMGV session, Post assessments will be conducted within 4 weeks of the final IMGV session.
  Patient report of physical function will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v2.0 Physical Function Short Form 4-a. This includes 4 questions assessing chores, ability to use stairs, walking, and running errands on a 5-point scale with end points of "without any difficulty" and "unable to do." Raw total scores range from 4-20, where a higher score correlates to a better outcome for physical function.
Change in Anxiety | Pre-assessments will be conducted within 4 weeks of the first IMGV session, Post assessments will be conducted within 4 weeks of the final IMGV session.
  Patient report of anxiety will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 Anxiety Short Form 4-a. This includes 4 questions assessing feeling fearful, ability to focus on anything other than anxiety, worries, and feeling uneasy in the past 7 days on a 5-point scale with end points of "never" and "always." Higher scores reflect more difficulty. Raw total scores range from 4-20, where a higher score correlates to a worse outcome for anxiety.
Change in Depression | Pre-assessments will be conducted within 4 weeks of the first IMGV session, Post assessments will be conducted within 4 weeks of the final IMGV session.
  Patient report of depression will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 - Emotional Distress-Depression - Short Form 4a. This includes 4 questions assessing feeling worthless, helpless, depressed, or hopeless in the past 7 days on a 5-point scale with end points of "never" and "always." Raw total scores range from 4-20, where a higher score correlates to a worse outcome for depression.
Change in Fatigue | Pre-assessments will be conducted within 4 weeks of the first IMGV session, Post assessments will be conducted within 4 weeks of the final IMGV session.
  Patient report of fatigue will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 -Fatigue - Short Form 4a. This includes 4 questions assessing feeling fatigued, had trouble starting things because of feeling tired, run-down, and fatigued on average in the past 7 days on a 5-point scale with end points of "not at all" and "very much." Raw total scores range from 4-20, where a higher score correlates to a worse outcome for fatigue.
Change in Sleep Disturbance | Pre-assessments will be conducted within 4 weeks of the first IMGV session, Post assessments will be conducted within 4 weeks of the final IMGV session.
  Patient report of sleep disturbance will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 -Sleep Disturbance - Short form 4a. This includes 4 questions assessing sleep quality, sleep was refreshing, problem with sleep, or difficulty falling asleep on average in the past 7 days on a 5-point scale with end points of "very poor" "very good" sleep quality and "not at all" and "very much" for all other questions. Raw total scores range from 4-20, where a higher score correlates to a worse outcome for sleep disturbance.
Change in Ability to Participate in Social Roles and Activities | Pre-assessments will be conducted within 4 weeks of the first IMGV session, Post assessments will be conducted within 4 weeks of the final IMGV session.
  Patient report of ability to participate in social roles and activities will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v2.0 - Ability to Participate in Social Roles and Activities- Short Form 4a. This includes 4 questions assessing trouble doing regular leisure activities with others, trouble doing family activities, trouble doing usual activities at work, and trouble doing activities with friend on a 5-point scale with end points of "never" and "always." Raw total scores range from 4-20, where a higher score correlates to a better outcome for ability to participate in social roles and activities.
Change in Pain Interference | Pre-assessments will be conducted within 4 weeks of the first IMGV session, Post assessments will be conducted within 4 weeks of the final IMGV session.
  Patient report of pain interference will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.1 - Pain Interference - Short Form 4a. This includes 4 questions assessing pain interfering with day to day activities, work around the home, ability to participate in social activities, and household chores in the past 7 days on a 5-point scale with end points of "not at all" and "very much." Higher scores reflect more difficulty. Raw total scores range from 4-20, where a higher score correlates to a better outcome for pain interference.
Change in Pain Intensity | Pre-assessments will be conducted within 4 weeks of the first IMGV session, Post assessments will be conducted within 4 weeks of the final IMGV session.
  Change in pain intensity will be measured before and after participation in the IMGV and assessed by the Pain Intensity sub-scale of the PROMIS-29 instrument. Pain intensity rating: 1 item from the Patient Reported Outcomes Measurement Information System (PROMIS), with pain intensity rated on 0-10 scale with lower values indicating less pain, or better outcome.
Change in Pain Medication Use | Assessments will be conducted within 4 weeks of the final IMGV session.
  Total pain medication use will be compared through data from the electronic health record (comparing medications listed before initiating and after participation in IMGV).

CONTACTS AND LOCATIONS:
Overall Officials: Isabel J Roth, DrPH, MS, Principal Investigator — University of North Carolina at Chapel Hill School of Medicine
Locations (1):
- University of North Carolina at Chapel Hill School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.